CLINICAL TRIAL: NCT04377152
Title: Expanded Access: 68Gallium-PSMA-11 for PET Imaging of Prostate Cancer
Brief Title: Expanded Access 68Gallium-PSMA-11 PET for Prostate Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Other Study IDs: EA-HOPE20200129; 20-30046 (Other: University of California, San Francisco)
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer; Prostate; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: 68Gallium-PSMA-11 — PSMA-11 Ga 68 Injection is a positron emitting radiopharmaceutical containing radioactive 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC (PSMA-11), which is used for diagnostic purposes in conjunction with Positron Emission Tomography (PET).
  Other Names: PSMA-HBED-CC
Procedure: Positron Emission Tomography (PET) — A PET scan is an imaging test that helps reveal how your tissues and organs are functioning using a radioactive drug (tracer) to show this activity
  Other Names: PET; PET Scan

SUMMARY:
This expanded access protocol provides eligible participants with investigational 68Ga-PSMA-11 PET imaging to detect and localize prostate cancer for initial and subsequent treatment strategy.

ELIGIBILITY:
Biochemical recurrent and pre-prostatectomy staging participants will be eligible and must meet the following criteria:

Inclusion Criteria:

1. Age ≥ 18 years
2. Histopathologically confirmed or biopsy proven prostate adenocarcinoma.
3. Concern for metastatic disease in one of the following settings:

   1. Initial staging with intermediate to high risk prostate cancer.
   2. Biochemical recurrence after initial therapy.
4. Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States